CLINICAL TRIAL: NCT06074744
Title: Subsartorial Saphenous Nerve Block (SSNB) Versus Femoral Nerve Block (FNB) in Primary Total Knee Arthroplasty (TKA) Combined With Infiltration Between Popliteal Artery and Capsule of the Knee (IPACK) - Where Are the Benefits?
Brief Title: Subsartorial Nerve Block and Femoral Nerve Block in Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Judith Bering, Principal Investigator, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSNB2023
Record Dates: First submitted 2023-08-23; First posted 2023-10-10 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Joint Diseases; Joint Pain
Keywords: Subsartorial Saphenous Nerve Block (SSNB); Femoral Nerve Block (FNB); Total Knee Arthroplasty (TKA)
MeSH Terms: conditions — Joint Diseases; Arthralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomization by sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: SSNB + IPACK (group 1) (Active Comparator): Subsartorial Nerve Block:
  * 15ml bupivacaine 0.5% + clonidine 1mcg/kg for prolongation of the block effect
  * anatomic landmarks: proximal adductor channel, intersection of the medial borders of the sartorius muscle and the adductor longus, guided by ultrasound control
  * no patch to puncture site to not jeopardise the surgeon's blinding
  * IPACK: 15ml bupivacaine 0.5% after completion of the femoral preparation
  Interventions: Other: SSNB + IPACK
- Control group: FNB + IPACK (group 2) (Active Comparator): Femoral Nerve Block:
  * 15ml bupivacaine 0.5% + clonidine 1mcg/kg for prolongation of the block effect
  * anatomic landmarks: lateral to the femoral artery,level of the femoral crease (proximal to the vascular outlet of the deep artery of the thigh), femoral nerve lies on the surface of the iliopsoas muscle and is covered by the fascia iliaca, guided by ultrasound control
  * no patch to puncture site to not jeopardise the surgeon's blinding
  * IPACK: 15ml bupivacaine 0.5% after completion of the femoral preparation
  Interventions: Other: FNB + IPACK

INTERVENTIONS:
Other: SSNB + IPACK — already included in arm/group description
  Other Names: Subsartorial Nerve Block
  Arms: Intervention group: SSNB + IPACK (group 1)
Other: FNB + IPACK — already included in arm/group description
  Other Names: Femoral Nerve Block
  Arms: Control group: FNB + IPACK (group 2)

SUMMARY:
The goal of this clinical trial is to compare two different types of nerve blocks in patients undergoing surgery for primary Total Knee Arthroplasty. The main question aim to answer is:

- is there a benefit in functional muscle power output of the leg?

Participants will be randomized into either the intervention group or the control group and:

* receive Subsartorial Saphenous Nerve Block (SSNB) + IPACK in intervention group (group 1)
* receive Femoral Nerve Block (FNB) + IPACK in control group (group 2)

Researchers will compare the 2 groups to see if there are differences in :

* functional muscle power output of the leg?
* muscle function, mobility, clinical and radiological results, ROM, pain control (NRS), opioid consumption, length of hospital stay, patient satisfaction, mobility, reduction of costs?

DETAILED DESCRIPTION:
Prospective, randomized, double-blinded, single-center, controlled clinical trial with intervention group (SSNB + IPACK, group 1) and control group (FNB + IPACK, group 2), randomization by sealed envelopes.

The number of participants will be 72 per group, calculated based on a sample size calculator program.

The 3 surgeons will be blinded as well as the patients regarding the nerve block they will receive.

We will explain to the patients how both the blocks will be carried out, that 1 block will be located "higher on the leg" and 1 "lower on the leg". The nerve blocks will be carried out by a well-trained anaesthesiologist following standard procedures preoperative.

The IPACK will be applied by the surgeons intraoperative, following a standard protocol. The used implant for all patients will be the cemented ATTUNE™ Primary Knee System® (DePuySynthes Johnson&Johnson).

Every patient will wear a brace fixed in full extension after surgery for the first 24 hours. Postoperative all patients will receive a standard set of adequate analgesics.

The postoperative rehabilitation program will follow our well-established physiotherapy scheme.

Performed assessments:

* Range of motion (ROM)
* medical history
* physical examinations
* radiologic controls
* adverse events
* falls during hospital stay (standard protocol)
* pain assessment (numeric rating scale)
* Questionnaires (EQ-5D-5L und Oxford Knee Score) will be filled in by the patients
* Functional assessment: Cycle sprint test one a specially instrumented indoor bike (Verve Info Tec PTY LTD) fit with an instrumented crank (InfoCrank Power Meter, Verve Cycling, West Perth, Australia)
* Functional assessment: Manual muscle testing (MMT)
* Functional assessment: Timed up and go test (TUG)

Superiority analysis using a two sample t-test, significance level 0.05, power 80%.

Data will be stored electronically in the data base (RedCap). In case of missing data there will always be attempts to obtain these data afterwards (contacting the patients by phone). Further on statistical analysis is performed.

Dropouts, before the 6 weeks follow-up, will be replaced by recruitment of new subjects.

For quality assurance the sponsor, the Ethics Committee or an independent trial monitor may visit the research sites.

ELIGIBILITY:
Inclusion criteria:

* age > 18yrs
* primary TKA
* BMI 35kg/m2 or less
* able to give informed consent as documented by signature
* clinical history without any contraindications for the planned intervention

Exclusion criteria:

* age < 18 years
* revision-TKA
* BMI >35kg/m2
* absent contact information
* inability or contraindications to undergo the investigated intervention (TKA, FNB, SSNB), - clinically significant concomitant diseases
* pregnancy
* inability to follow the procedures and follow-up procedures of the study (e.g. due to language problems, psychological disorders, dementia, living abroad, etc.
* withdrawal from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Functional muscle power output of the leg | preoperative, 6 weeks, 12 weeks, 1 year after surgery
  Cycle sprint test measuring maximum lower limb muscle power in Watts (W) from 3 times 10-second maximal efforts (higher values better)

SECONDARY OUTCOMES:
Muscle strength | preoperative, 48 hours after surgery, day of discharge (7+/- 2 days postoperative), 6 weeks, 12 weeks, 1 year after surgery
  Manual muscle testing (MMT) as a standardized measuring tool to assess quadriceps muscle strength using a numeric score 0-5 (Daniels and Worthingham Scale): patient in sitting position in 20 degree knee flexion is asked to extend the knee actively against resistance proximal to the ankle (higher values better)
Mobility | preoperative, 48 hours after surgery, day of discharge (7+/- 2 days postoperative), 6 weeks, 12 weeks1 year after surgery
  Timed up and go test (TUG): standardized measuring tool, the patient is timed while they rise from an arm chair (approximate seat height 46 cm), walk at a comfortable and safe pace to a line on the floor 3 metres away, turn and walk back to the chair and sit down again (in seconds) (lower values better)
Clinical results | preoperative, day of discharge (7+/- 2 days postoperative), 6, 12 weeks, 1 year after surgery
  redness, swelling, hyperthermia, wound/scar, range of motion, stability, adverse events
Radiological results | preoperative(1-3), day 1 after surgery(1), 6 weeks(1-2), 1 year after surgery(1-3)
  x-rays ap and lateral view(1), patella(2), whole leg axis(3)
Pain control | before surgery, twice daily on the ward (except first 6 hours: hourly), day of discharge (7+/- 2 days postoperative), 6 weeks, 12 weeks, 1 year after surgery
  numeric rating scale 0-10 (lower values better)
Opioid consumption | before surgery, during hospital stay, day of discharge (7+/- 2 days postoperative), 6 weeks, 12 weeks, 1 year after surgery
  documentation of administered drugs including name of drug, dosage, frequency of use
Length of hospital stay | before surgery, during hospital stay, day of discharge (7+/- 2 days postoperative), 6 weeks, 12 weeks, 1 year after surgery
  documentation of days in hospital
Patient satisfaction 1 | preoperative, 6 weeks, 12 weeks, 1 year after surgery
  Questionnaire (Oxford Knee Score) 12-60 points (lower values better)
Patient satisfaction 2 | preoperative, 6 weeks, 12 weeks, 1 year after surgery
  Questionnaire (EQ-5D-5L) 5 questions with 5 answers each (lower values better) including EQ-VAS 0-100 (higher values better)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Bering, Dr. med., Principal Investigator — Luzerner Kantonsspital Luzern
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Declaration of Helsinki, Version October 2013
- [Background] International Conference on Harmonization (ICH) E6(R2) Guideline for Good Clinical Practice
- [Background] International Conference on Harmonization (ICH, 1997) E8 Guideline: General Considerations for Clinical Trials
- [Background] Implantatregister SIRIS Hüfte und Knie: Kurzfassung - SIRIS Report 2022
- [Background] Bundesamt für Statistik, Schweiz
- [Background] Grosu I, Lavand'homme P, Thienpont E. Pain after knee arthroplasty: an unresolved issue. Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1744-58. doi: 10.1007/s00167-013-2750-2. Epub 2013 Nov 8. PMID 24201900
- [Background] Burket LW, Greenberg MS, Glick M. Burkett's Textbook of Oral Medicine. 10th ed. Philadelphia, PA: Lippincott
- [Background] Winnie AP, Ramamurthy S, Durrani Z. The inguinal paravascular technic of lumbar plexus anesthesia: the "3-in-1 block". Anesth Analg. 1973 Nov-Dec;52(6):989-96. No abstract available. PMID 4796576
- [Background] Tierney E, Lewis G, Hurtig JB, Johnson D. Femoral nerve block with bupivacaine 0.25 per cent for postoperative analgesia after open knee surgery. Can J Anaesth. 1987 Sep;34(5):455-8. doi: 10.1007/BF03014348. PMID 3664912
- [Background] Rosenblatt RM. Continuous femoral anesthesia for lower extremity surgery. Anesth Analg. 1980 Aug;59(8):631-2. No abstract available. PMID 7190803
- [Background] Edwards ND, Wright EM. Continuous low-dose 3-in-1 nerve blockade for postoperative pain relief after total knee replacement. Anesth Analg. 1992 Aug;75(2):265-7. doi: 10.1213/00000539-199208000-00020. PMID 1632541
- [Background] Ma HH, Chou TA, Tsai SW, Chen CF, Wu PK, Chen WM. The efficacy of continuous versus single-injection femoral nerve block in Total knee Arthroplasty: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2020 Feb 24;21(1):121. doi: 10.1186/s12891-020-3148-1. PMID 32093655
- [Background] Atkinson HD, Hamid I, Gupte CM, Russell RC, Handy JM. Postoperative fall after the use of the 3-in-1 femoral nerve block for knee surgery: a report of four cases. J Orthop Surg (Hong Kong). 2008 Dec;16(3):381-4. doi: 10.1177/230949900801600324. PMID 19126912
- [Background] Sharma S, Iorio R, Specht LM, Davies-Lepie S, Healy WL. Complications of femoral nerve block for total knee arthroplasty. Clin Orthop Relat Res. 2010 Jan;468(1):135-40. doi: 10.1007/s11999-009-1025-1. Epub 2009 Aug 13. PMID 19680735
- [Background] Feibel RJ, Dervin GF, Kim PR, Beaule PE. Major complications associated with femoral nerve catheters for knee arthroplasty: a word of caution. J Arthroplasty. 2009 Sep;24(6 Suppl):132-7. doi: 10.1016/j.arth.2009.04.008. Epub 2009 Jun 24. PMID 19553071
- [Background] Runner RP, Boden SA, Godfrey WS, Premkumar A, Samady H, Gottschalk MB, Xerogeanes JW. Quadriceps Strength Deficits After a Femoral Nerve Block Versus Adductor Canal Block for Anterior Cruciate Ligament Reconstruction: A Prospective, Single-Blinded, Randomized Trial. Orthop J Sports Med. 2018 Sep 26;6(9):2325967118797990. doi: 10.1177/2325967118797990. eCollection 2018 Sep. PMID 30276220
- [Background] Luo TD, Ashraf A, Dahm DL, Stuart MJ, McIntosh AL. Femoral nerve block is associated with persistent strength deficits at 6 months after anterior cruciate ligament reconstruction in pediatric and adolescent patients. Am J Sports Med. 2015 Feb;43(2):331-6. doi: 10.1177/0363546514559823. Epub 2014 Dec 2. PMID 25466410
- [Background] Everhart JS, Hughes L, Abouljoud MM, Swank K, Lewis C, Flanigan DC. Femoral nerve block at time of ACL reconstruction causes lasting quadriceps strength deficits and may increase short-term risk of re-injury. Knee Surg Sports Traumatol Arthrosc. 2020 Jun;28(6):1894-1900. doi: 10.1007/s00167-019-05628-7. Epub 2019 Jul 17. PMID 31317214
- [Background] Brull R, McCartney CJ, Chan VW, El-Beheiry H. Neurological complications after regional anesthesia: contemporary estimates of risk. Anesth Analg. 2007 Apr;104(4):965-74. doi: 10.1213/01.ane.0000258740.17193.ec. PMID 17377115
- [Background] van der Wal M, Lang SA, Yip RW. Transsartorial approach for saphenous nerve block. Can J Anaesth. 1993 Jun;40(6):542-6. doi: 10.1007/BF03009739. PMID 8403121
- [Background] Mansour NY. Sub-sartorial saphenous nerve block with the aid of nerve stimulator. Reg Anesth. 1993 Jul-Aug;18(4):266-8. No abstract available. PMID 8398966
- [Background] Abdallah FW, Whelan DB, Chan VW, Prasad GA, Endersby RV, Theodoropolous J, Oldfield S, Oh J, Brull R. Adductor Canal Block Provides Noninferior Analgesia and Superior Quadriceps Strength Compared with Femoral Nerve Block in Anterior Cruciate Ligament Reconstruction. Anesthesiology. 2016 May;124(5):1053-64. doi: 10.1097/ALN.0000000000001045. PMID 26938989
- [Background] Maye A, Hurley E, Jamal M, Curley G. Adductor canal block versus femoral nerve block in total knee arthroplasty: a Meta-Analysis of randomized control trials. ESRA 2019 19-0449
- [Background] Fan Chiang YH, Wang MT, Chan SM, Chen SY, Wang ML, Hou JD, Tsai HC, Lin JA. Motor-Sparing Effect of Adductor Canal Block for Knee Analgesia: An Updated Review and a Subgroup Analysis of Randomized Controlled Trials Based on a Corrected Classification System. Healthcare (Basel). 2023 Jan 10;11(2):210. doi: 10.3390/healthcare11020210. PMID 36673579
- [Background] Hasabo EA, Assar A, Mahmoud MM, Abdalrahman HA, Ibrahim EA, Hasanin MA, Emam AK, AbdelQadir YH, AbdelAzim AA, Ali AS. Adductor canal block versus femoral nerve block for pain control after total knee arthroplasty: A systematic review and Meta-analysis. Medicine (Baltimore). 2022 Aug 26;101(34):e30110. doi: 10.1097/MD.0000000000030110. PMID 36042669
- [Background] Sinha S, Abras J, Sivasenthil D. Use of ultrasound guided popliteal fossa infiltration to control pain after total knee arthroplasty: a prospective randomized observer-blinded study. ASRA 37th Annual Regional Anesthesia Meeting and Workshops; March 15-18, San Diego, CA, 2012
- [Background] Chan E, Howle R, Onwochei D, Desai N. Infiltration between the popliteal artery and the capsule of the knee (IPACK) block in knee surgery: a narrative review. Reg Anesth Pain Med. 2021 Sep;46(9):784-805. doi: 10.1136/rapm-2021-102681. Epub 2021 May 14. PMID 33990439
- [Background] Guo J, Hou M, Shi G, Bai N, Huo M. iPACK block (local anesthetic infiltration of the interspace between the popliteal artery and the posterior knee capsule) added to the adductor canal blocks versus the adductor canal blocks in the pain management after total knee arthroplasty: a systematic review and meta-analysis. J Orthop Surg Res. 2022 Aug 12;17(1):387. doi: 10.1186/s13018-022-03272-5. PMID 35962410
- [Background] Mou P, Wang D, Tang XM, Zeng WN, Zeng Y, Yang J, Zhou ZK. Adductor Canal Block Combined With IPACK Block for Postoperative Analgesia and Function Recovery Following Total Knee Arthroplasty: A Prospective, Double-Blind, Randomized Controlled Study. J Arthroplasty. 2022 Feb;37(2):259-266. doi: 10.1016/j.arth.2021.10.004. Epub 2021 Oct 13. PMID 34653576
- [Background] Hurworth M, Evans JM, Gibbons R, Mackie KE, Edmondston SJ. Cycle Sprint Test for the Evaluation of Lower Limb Muscle Power After Total Knee Arthroplasty: A Proof-of-Concept Study. Arthroplast Today. 2021 Jun 15;9:118-121. doi: 10.1016/j.artd.2021.05.007. eCollection 2021 Jun. PMID 34189216
- [Background] Wright, W. Muscle training in the treatment of infantile paralysis. Boston Med. Surg. J. 1912, 167, 567-574
- [Background] Li D, Alqwbani M, Wang Q, Liao R, Yang J, Kang P. Efficacy of Adductor Canal Block Combined With Additional Analgesic Methods for Postoperative Analgesia in Total Knee Arthroplasty: A Prospective, Double-Blind, Randomized Controlled Study. J Arthroplasty. 2020 Dec;35(12):3554-3562. doi: 10.1016/j.arth.2020.06.060. Epub 2020 Jun 24. PMID 32680754
- [Background] Collins NJ, Misra D, Felson DT, Crossley KM, Roos EM. Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S208-28. doi: 10.1002/acr.20632. No abstract available. PMID 22588746
- [Background] EQ-5D-3L Manual Guide. Euroquol.org. 2021 [cited 28 March 2021]. vailable from: https://euroquol.org/wp-content/uploads/2019/10/EQ-5D-3L-User-Guide_version-6.0.pd
- [Background] Lam CLK, Tse ETY, Wong CKH, Lam JSM, Chen SS, Bedford LE, Cheung JPY, Or CK, Kind P. A pilot study on the validity and psychometric properties of the electronic EQ-5D-5L in routine clinical practice. Health Qual Life Outcomes. 2021 Dec 18;19(1):266. doi: 10.1186/s12955-021-01898-3. PMID 34922564
- [Background] Stocks GW, Odoemene M, Gex J, Vidal EA, Sawyer K, Jones SL, Thompson B, Laughlin MS. Quadriceps Strain and TKA: Contribution of the Tourniquet and Intramedullary Rod to Postoperative Thigh Pain: A Randomized Controlled Trial. J Bone Joint Surg Am. 2023 Mar 15;105(6):455-461. doi: 10.2106/JBJS.22.00703. Epub 2023 Jan 9. PMID 36728455
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Barry E, Galvin R, Keogh C, Horgan F, Fahey T. Is the Timed Up and Go test a useful predictor of risk of falls in community dwelling older adults: a systematic review and meta-analysis. BMC Geriatr. 2014 Feb 1;14:14. doi: 10.1186/1471-2318-14-14. PMID 24484314
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Common Terminology Criteria for Adverse Events (CTCAE) https://www.eortc.be/services/doc/ctc/CTCAE_4.03_2010-06-14_QuickReference_5x7.pdf
- [Background] Federal Act on Data Protection (FADP) https://www.admin.ch/opc/en/classified-compilation/19920153/index.html
- [Background] Human Research Act (HRA) https://www.admin.ch/opc/de/classified-compilation/20061313/index.html
- [Background] International Conference on Harmonization (ICH) E2A Clinical Safety Data Management: Definitions and Standards for Expedited Reporting http://www.ema.europa.eu/docs/en_GB/document_library/Scientific_guideline/2009/09/WC500002749.pdf
- [Background] Ordinance on Clinical Trials in Human Research (ClinO) https://www.admin.ch/opc/de/classified-compilation/20121176/index.html